CLINICAL TRIAL: NCT02485418
Title: Low- Dose Propofol Infusion as an Abortive Treatment for Migraine Headaches in Pediatric Patients
Acronym: Propofol2014
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Deryk Walsh, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 042014-002
Record Dates: First submitted 2015-06-04; First posted 2015-06-30 (Estimated); Results first posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Propofol infusion (Experimental): All subjects will be treated with an intravenous propofol infusion at the following escalating rate schedule:
  20 mcg/kg/min for 10 minutes, followed by an increase to 30 mcg/kg/min for 10 minutes and then by an increase to 40 mcg/kg/min for 40 minutes
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Intravenous propofol infusion at 20 mcg/kg/min for 10 minutes, followed by an increase to 30 mcg/kg/min for 10 minutes and then by an increase to 40 mcg/kg/min for 40 minutes.

SUMMARY:
Propofol has been used in adult populations to treat migraines as an abortive agent. Investigators plan to investigate its efficacy as an abortive agent in the pediatric population when administered as a safe low-dose infusion. Goals of the study are to:

1. Evaluate efficacy of low-dose propofol infusion as an abortive agent in pediatric migraine headaches
2. Evaluate effective and safe dosing limits in pediatric populations
3. Evaluate duration of effect reached from a low-dose propofol infusion as an abortive agent

Endpoints for the study will be:

1. Number of enrolled patients
2. Safety endpoints reached, including: cardiopulmonary depression, excessive somnolence Risks of the study are minimal due to the use of sub-anesthetic dosing of propofol under the guidance and supervision of a board certified pediatric anesthesiologist with the appropriate monitoring equipment and readily available emergency equipment. Investigators hope to demonstrate more rapid improvement and decreased side-effect as compared to standard care.

DETAILED DESCRIPTION:
The aim of this prospective study is to evaluate the efficacy and safety of propofol administration in a hospital setting, as an abortive medication for children aged 7-18 with migraines.

Primary outcome:

Based on the adult and the limited pediatric data available we hypothesize that propofol infusion in sub anesthetic dose, will result in either complete resolution or improve the headache pain scores by 50% from the baseline pain scores. Patients will be assessed with a 0-10 Numeric Pain Rating Scale.

Secondary outcomes:

* Time to beginning of effect (from the beginning of the propofol infusion till first improvement in pain score noted)
* Duration of effect (from the end of propofol administration till discharge criteria are meet or if treatment is ineffective, till start of new therapy)
* Total propofol dose based on weight.

Prior to initiation of DHE infusion, the subjects will receive sub-anesthetic doses of propofol infusion:

20 mcg/kg/min for 10 minutes, followed by an increase to 30 mcg/kg/min for 10 minutes and then by an increase to 40 mcg/kg/min for 40 minutes. The propofol infusion will be terminated if:

* The patient has no pain, or greater than 50% reduction in pain scores as compared to the pretreatment pain score
* After completing 40 minutes of propofol infusion at 40 mcg/kg/min irrespective of the pain score
* If the anesthesiologist feels cardio-pulmonary depression, airway obstruction or over sedation (Ramsay Sedation Score greater than 3)has occurred

If the propofol infusion is effective in resolving headache symptoms, then subjects will be monitored for at least 30 minutes after termination of infusion. Outpatient subjects would then be discharged home; inpatient subjects would resume standard care treatment.

If propofol infusion is not successful in resolving headache, then the subjects will proceed with DHE infusion per standard of care. If the subject still has no relief, the study investigators will discuss further options with the subject and parents, including hospital admission for further therapy for outpatient subjects.

For all subjects who receive propofol infusion, follow-up will occur at 24 and 48 hours via phone call to evaluate headache status and recover information on headache symptoms and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of migraine headache per ICHD - 3 (International Classification of Headache Disorders)
* The subjects will have a history of migraine headaches with a presentation consistent with presentations of their headaches in the past with no indication for further investigation for secondary causes of his/her headache
* Documented pain score greater than or equal to 6 on a 0-10 Numeric Pain Rating Scale
* Current migraine has a greater than 24 hours duration with a current pain score of 6 or greater on a 0-10 Numeric Pain Rating Scale
* Subjects will be scheduled for DHE infusion therapy for treatment of migraines per standard medical care
* Patients age 7-18 years old
* Gender: both male and female
* Appropriate fasting interval as per ASA guidelines

Exclusion Criteria:

* No long acting triptan therapy within 24 hours
* No shorter acting triptan therapy within 6 hours
* No ergot alkaloid derivatives within the last 24 hours
* No opioid within 2 hours
* No NSAID or acetaminophen within 1 hour of infusion
* Use of sedative medications within 6 hours of infusion, including opioids, benzodiazepines, barbiturates
* Headache not consistent with subject's headache history needing further work-up
* Headache duration less than 24 hours
* Subjects in which an intravenous line could not be secured
* Subjects with history of significant reflux or hiatal hernia
* Subjects with history of significant cardio pulmonary disorders
* Patient not fasting as per ASA guidelines

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deryk Walsh, MD, Principal Investigator — Children's Medical Center Dallas
Locations (1):
- Children's Health Children's Medical Center Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two headache clinic populations
Pre-assignment Details: Forty patients met criteria and were enrolled.
Groups:
- Propofol Infusion: All subjects will be treated with an intravenous propofol infusion at the following escalating rate schedule:
  20 mcg/kg/min for 10 minutes, followed by an increase to 30 mcg/kg/min for 10 minutes and then by an increase to 40 mcg/kg/min for 40 minutes
  Propofol: Intravenous propofol infusion at 20 mcg/kg/min for 10 minutes, followed by an increase to 30 mcg/kg/min for 10 minutes and then by an increase to 40 mcg/kg/min for 40 minutes.
Period: Overall Study
Arm/Group | Propofol Infusion
Started | 40
Completed | 38
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: 40 patients screened and 2 patients excluded and baseline characteristics not included
Arm/Group | Propofol Infusion
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 38
Number of Participants [Count of Participants; unit: Participants] | 38

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Headache Pain Score
Description: Change in pain score on 0-10 Numeric Pain Rating Scale with 0 being no pain and 10 being severe pain. Subjects assessed at 10 minute intervals for the duration of the infusion with reporting of change from baseline to 60 minutes
Time Frame: Duration of propofol infusion (between 5 and 60 minutes)
Population: Per protocol, analysis of data based on patients completing 60 minute infusion of propofol
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Propofol Infusion
Number analyzed (Participants) | 40
score on a scale | -3.3 (2.5)

2. Secondary Outcome: NPRS Pain Scores at 24 and 48 Hours Post Infusion
Description: For subjects who experience a change in pain score or who report resolution from headache symptoms, duration of analgesia up to 48 hours after treatment,characterized by NPRS Pain scores on a scale of 0-10 with 0 being no pain and 10 being severe pain.
Time Frame: Assessments of NPRS Pain scores on a scale of 0-10 with 0 being no pain and 10 being severe pain at 24 and 48 hours after discharge from infusion
Measure: Mean (Standard Deviation); unit: Pain Score 0-10 scale
Arm/Group | Propofol Infusion
Number analyzed (Participants) | 38
Pain Score 0-10 scale
  Baseline | 7.5 (1.3)
  24 hours post infusion | 4.3 (2.6)
  48 hours post infusion | 3.4 (2.7)

3. Secondary Outcome: Total Propofol Dose
Description: Total dose of propofol administered (mg/kg)
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: mg/kg
Groups:
- Total Dose of Propofol Administered (mg/kg): Each patient enrolled received the protocol dosing of propofol as outlined. All patients received scheduled 2.1 mg/kg over 60 minutes as per protocol, except for one patient who was discontinued due to complete resolution of headache. Considered outlier.
Arm/Group | Total Dose of Propofol Administered (mg/kg)
Number analyzed (Participants) | 38
mg/kg | 2.1 (0)

ADVERSE EVENTS:
Time Frame: 48 hours
Description: Adverse events were collected by nursing at time of infusion and 24 and 48 hours post infusion by phone communication.
  All-Cause Mortality was not monitored/assessed.
Arm/Group | Propofol Infusion
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 1/38
Other Adverse Events (participants affected / at risk) | 2/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propofol Infusion (N=38)
emesis, abdominal pain & fever (Gastrointestinal disorders) | 1 (1) — patient with emesis, abdominal pain and fever at 24 hour follow-up. Patient seen in the ED 1 week prior to infusion with similar symptoms.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propofol Infusion (N=38)
nausea (Gastrointestinal disorders) | 2 (2) — Patients with nausea with peripheral intravenous line insertion, prior to infusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT02485418/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT02485418/SAP_001.pdf